CLINICAL TRIAL: NCT02069899
Title: A Multicenter Study for the Long-term Follow-up of HLH Patients Who Received Treatment With NI-0501, an Anti-interferon Gamma Monoclonal Antibody
Brief Title: A Study for Long-term Follow-up of Hemophagocytic Lymphohistiocytosis (HLH) Participants Who Received Treatment With Emapalumab (NI-0501), an Anti-interferon Gamma Monoclonal Antibody
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Seventh Framework Programme (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NI-0501-05
Record Dates: First submitted 2013-12-23; First posted 2014-02-24 (Estimated); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-05

CONDITIONS: Hemophagocytic Lymphohistiocytosis
Keywords: Hemophagocytic lymphohistiocytosis (HLH) previously treated with NI-0501; Emapalumab
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Emapalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (3):
- Enrolled-04 Cohort (Other): Participants enrolled in Study NI-0501-04 (NCT01818492) will be invited to participate for long-term follow-up for 1 year either after haematopoietic stem cell transplantation (HSCT) or after the last administration of emapalumab.
  In Study NI-0501-04, participants received emapalumab for 4 to 8 weeks. After the treatment period, participants could have undergone HSCT.
  Participants for whom an appropriate donor was not identified by Week 8, or in a case where HSCT will be delayed for reasons unrelated to the administration of emapalumab, can continue receiving treatment with emapalumab beyond the foreseen 8 weeks in the current study (NI-0501-05, NCT02069899) at the request of the investigator, providing a favorable benefit/risk assessment of treatment is established.
  The dose and timing was either carried forward from the last administered emapalumab dose as part of the parent protocol or an adjusted dose was administered, if necessary.
  Interventions: Drug: Emapalumab
- Enrolled-06 Cohort (No Intervention): All participants who received at least 1 dose of emapalumab and were monitored for at least 4 weeks after the last drug administration in Study NI-0501-06 (NCT03311854) will be invited to participate for long-term follow-up for 1 year after the last administration of emapalumab.
  Participants will not receive emapalumab in the current study (NI-0501-05, NCT02069899).
- Enrolled-CU Cohort (Other): In exceptional cases, at the spontaneous request of a treating physician, CU treatment will be granted to the participants who had exhausted all possible treatment options and who could not be enrolled in a clinical study. All participants who receive at least 1 dose of emapalumab under CU will be invited to participate for long-term follow-up for 1 year either after HSCT or after the last administration of emapalumab.
  Participants can continue treatment in the context of the current Study (NI-0501-05, NCT02069899) while stem cell donor search is ongoing, or if the investigator assesses that continuation of treatment is beneficial.
  Interventions: Drug: Emapalumab

INTERVENTIONS:
Drug: Emapalumab — Treatment with emapalumab is not planned for all enrolled participants. For participants who will continue receiving emapalumab in the context of this study (NI-0501-05), the dose and timing will be either carried forward from the last administered emapalumab dose as part of the parent study in which the participant was enrolled, or an adjusted dose will be administered, if necessary.
  Other Names: NI-0501
  Arms: Enrolled-04 Cohort; Enrolled-CU Cohort

SUMMARY:
International, multicenter, long-term, follow-up study that will enrol HLH participants who have received emapalumab in previous clinical trials, in the context of the clinical development program for emapalumab or under compassionate use (CU).

DETAILED DESCRIPTION:
The aim of this study is to monitor the long-term safety profile of emapalumab in participants who have previously received at least one dose of emapalumab, including survival time after the administration of emapalumab.

Moreover, the elimination profile of emapalumab and the immunogenicity will also be assessed.

Furthermore, safety, tolerability, efficacy, and pharmacokinetic (PK) profile of emapalumab will be closely monitored in the event that some participants, upon request of the treating physician, will receive emapalumab treatment in the follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Having received at least one dose of emapalumab.
* Having signed the Informed Consent by the participant or the participant's legal representative(s), as applicable, with the assent of participant who are legally capable of providing it.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (5):
  - Spectrum Health Helen Devos Children's Hospital, Grand Rapids, Michigan
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital - Division of Immunobiology, Cincinnati, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Texas Children's Cancer Center, Houston, Texas
- Hôpital Necker-Enfants Malades, Paris, France
- Italy (5):
  - Fondazione MBBM c/o Ospedale San Gerardo Clinica Pediatrica, Monza
  - Azienda Ospedaliera Padova, Padua
  - Ospedale Pediatrico Bambino Gesu - UO Reumatologia, Rome
  - Ospedale Pediatrico Bambino Gesu, Rome
  - Ospedale della Donna e del Bambino - U.O.C. Oncoematologia Pediatrica, Verona
- Spain (3):
  - Hospital Universitario Vall d'Hebron Servei de Hematologia i Oncologia, Barcelona
  - Sant Joan de Déu Hospital - Pediatric Rheumatology Department, Barcelona
  - Hospital Universitario Niño Jesús Servicio de Hemato-Oncología Pediátrica, Madrid
- United Kingdom (2):
  - UCL Institute of Child Health Great Ormond Street Hospital, London
  - Great Ormond Street Hospital - Department of Haematology, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jordan MB, Locatelli F, Allen C, Cesaro S, Rizzari C, Rao A, Degar B, Garrington T, Sevilla J, Putti MC, Fagioli F, Ahlmann M, Dapena Diaz JL, Henry M, Grom A, De Benedetti F, de Min C. Post-Transplant Outcomes of Children with Primary Hemophagocytic Lymphohistiocytosis Treated with Emapalumab.Transplant Cell Ther. 2021; 27(Supplement 3): S118.
- [Result] Laveille C, Jacqmin P, de Graaf K, de Min C. Population Pharmacokinetic Analysis of Emapalumab, a Fully Human, Anti-Interferon Gamma Monoclonal Antibody, in Children with Primary Hemophagocytic Lymphohistiocytosis. Blood 2020; 136 (Supplement 1): 20
- [Result] Locatelli F, Jordan MB, Allen C, Cesaro S, Rizzari C, Rao A, Degar B, Garrington TP, Sevilla J, Putti MC, Fagioli F, Ahlmann M, Dapena Diaz JL, Henry M, De Benedetti F, Grom A, Lapeyre G, Jacqmin P, Ballabio M, de Min C. Emapalumab in Children with Primary Hemophagocytic Lymphohistiocytosis. N Engl J Med. 2020 May 7;382(19):1811-1822. doi: 10.1056/NEJMoa1911326. PMID 32374962
- [Derived] Brossard P, Laveille C. Population Pharmacokinetics of the Anti-Interferon-Gamma Monoclonal Antibody Emapalumab: An Updated Analysis. Rheumatol Ther. 2024 Jun;11(3):869-880. doi: 10.1007/s40744-024-00669-y. Epub 2024 Apr 25. PMID 38662147
- [Derived] De Benedetti F, Grom AA, Brogan PA, Bracaglia C, Pardeo M, Marucci G, Eleftheriou D, Papadopoulou C, Schulert GS, Quartier P, Anton J, Laveille C, Frederiksen R, Asnaghi V, Ballabio M, Jacqmin P, de Min C. Efficacy and safety of emapalumab in macrophage activation syndrome. Ann Rheum Dis. 2023 Jun;82(6):857-865. doi: 10.1136/ard-2022-223739. Epub 2023 Mar 31. PMID 37001971

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with hemophagocytic lymphohistiocytosis (HLH) who had received at least 1 dose of emapalumab in the context of a previous emapalumab clinical study (Study NI-0501-04 [NCT01818492] or Study NI-0501-06 [NCT03311854]) in which no long-term follow-up was planned, and participants who received emapalumab through a compassionate use (CU) were enrolled in the current study (NI-0501-05, NCT02069899).
Groups:
- Enrolled-04 Cohort: Participants enrolled in Study NI-0501-04 were invited to participate for long-term follow-up for 1 year either after haematopoietic stem cell transplantation (HSCT) or after the last administration of emapalumab.
  In Study NI-0501-04, participants received emapalumab for 4 to 8 weeks. After the treatment period, participants could have undergone HSCT.
  For participants for whom an appropriate donor was not identified by Week 8, or in a case where HSCT was delayed for reasons unrelated to the administration of emapalumab, they could continue receiving treatment with emapalumab beyond the foreseen 8 weeks in the current study (NI-0501-05) at the request of the investigator, providing a favorable benefit/risk assessment of treatment was established.
  Treatment with emapalumab was not planned for all enrolled participants. For participants who continued receiving emapalumab in the context of this study (NI-0501-05), the dose and timing was either carried forward from the last administered emapalumab dose as part of the parent study in which the participant was enrolled, or an adjusted dose was administered, if necessary.
- Enrolled-06 Cohort: All participants who received at least 1 dose of emapalumab and were monitored for at least 4 weeks after the last drug administration in Study NI-0501-06 were invited to participate for long-term follow-up for 1 year after the last administration of emapalumab.
  Participants did not receive emapalumab in the current study (NI-0501-05).
- Enrolled-CU Cohort: In exceptional cases, at the spontaneous request of a treating physician, CU treatment was granted to the participants who had exhausted all possible treatment options and who could not be enrolled in a clinical study. All participants who received at least 1 dose of emapalumab were invited to participate for long-term follow-up for 1 year either after HSCT or after the last administration of emapalumab.
  Participants could have continued treatment in the context of the current Study (NI-0501-05) while stem cell donor search was ongoing, or if the investigator assessed that continuation of treatment was beneficial.
Period: Overall Study
Arm/Group | Enrolled-04 Cohort | Enrolled-06 Cohort | Enrolled-CU Cohort
Started | 37 | 14 | 7
Treated in Current Study | 22 | 0 | 5
Completed | 24 | 13 | 4
Not Completed | 13 | 1 | 3
Not completed — Adverse Event | 6 | 0 | 1
Not completed — Withdrawal by Participant | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Other | 4 | 0 | 0
Not completed — Participant could not travel to the study site due to Covid restrictions | 0 | 1 | 0
Not completed — Participant was withdrawn to receive emapalumab again in CU and then subsequently died | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who previously received treatment in a parent study (NI-0501-04 or NI-0501-06) or under compassionate use and who provided informed consent for participation in Study NI-0501-05.
Groups:
- Enrolled-04 Cohort: Participants enrolled in Study NI-0501-04 were invited to participate for long-term follow-up for 1 year either after HSCT or after the last administration of emapalumab.
  In Study NI-0501-04, participants received emapalumab for 4 to 8 weeks. After the treatment period, participants could have undergone HSCT.
  For participants for whom an appropriate donor was not identified by Week 8, or in a case where HSCT was delayed for reasons unrelated to the administration of emapalumab, they could continue receiving treatment with emapalumab beyond the foreseen 8 weeks in the current study (NI-0501-05) at the request of the investigator, providing a favorable benefit/risk assessment of treatment was established.
  Treatment with emapalumab was not planned for all enrolled participants. For participants who continued receiving emapalumab in the context of this study (NI-0501-05), the dose and timing was either carried forward from the last administered emapalumab dose as part of the parent study in which the participant was enrolled, or an adjusted dose was administered, if necessary.
- Total: Total of all reporting groups
Arm/Group | Enrolled-04 Cohort | Enrolled-06 Cohort | Enrolled-CU Cohort | Total
Number analyzed (Participants) | 37 | 14 | 7 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37 | 13 | 7 | 57
  Between 18 and 65 years | 0 | 1 | 0 | 1
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 4 | 33
  Male | 18 | 4 | 3 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Caucasian | 27 | 11 | 5 | 43
  Race: Asian | 4 | 0 | 1 | 5
  Race: Black/African descent | 3 | 2 | 1 | 6
  Race: Other | 3 | 0 | 0 | 3
  Race: Not collected/Missing | 0 | 1 | 0 | 1
Ethnicity [Count of Participants; unit: Participants] — Population: Ethnicity not collected

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Event (AE)
Description: Adverse events were defined as any undesirable experience occurring in a participant during the study, whether or not considered related to emapalumab.
Time Frame: From the date of enrollment in this study up to 1 year either after HSCT or after the last administration of emapalumab (maximum duration: 639 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled-04 Cohort | Enrolled-06 Cohort | Enrolled-CU Cohort
Number analyzed (Participants) | 37 | 14 | 7
Participants | 37 | 12 | 7

2. Secondary Outcome: Cumulative Duration of Response (Enrolled-04 Cohort)
Description: Cumulative duration of response: total number of days in response from 1st achievement of overall response until HSCT or last treatment date if the participant did not undergo HSCT. Overall response: achievement of either Complete (CR) or Partial Response (PR), or HLH Improvement (HI).
  CR: no fever, normal spleen size, no cytopenia (absolute neutrophil count [ANC] ≥1.0 x 10^9/L and platelet count ≥ 100 x 10^9/L), no hyperferritinemia (serum ferritin <2000 μg/L), no coagulopathy (normal D-dimer and/or fibrinogen >150 mg/dL), no neurological and cerebrospinal fluid [CSF] abnormalities attributed to HLH, no sustained worsening of soluble cluster of differentiation (CD) 25.
  PR: at least 3 HLH clinical and laboratory criteria (including central nervous system [CNS] abnormalities) met the CR criteria, no progression of other aspects of HLH disease pathology.
  HI: improvement (>50% change from baseline) of at least 3 HLH clinical and laboratory abnormalities (including CNS involvement).
Time Frame: From 1st achievement of overall response until HSCT or last treatment date if participant did not undergo HSCT (maximum 250 days)
Population: Enrolled-04 population included participants previously enrolled and treated in Study NI-0501-04 (participants with primary HLH) who provided informed consent for participation in Study NI-0501-05 and who had at least 1 response.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Enrolled-04 Cohort
Number analyzed (Participants) | 36
days | 70.7 (56.35)

3. Secondary Outcome: Duration of First Response (Enrolled-06 Cohort)
Description: Duration of first response was defined as the number of days between first date of response and first date of loss of response or death. Response was defined as macrophage activation syndrome (MAS) remission, which was resolution of clinical signs and symptoms according to the Investigator (MAS clinical signs and symptoms score ≤ 1) and normalization of laboratory parameters relevant to MAS as follows: white blood cells (WBC) and platelet count above the upper limit of normal (LLN), Lactate dehydrogenase < 1.5 × lower limit of normal (ULN), aspartate aminotransferase/alanine aminotransferase <1.5 × ULN, fibrinogen > 100 mg/dL, ferritin level decreased by at least 80% from values at screening or baseline (whichever was higher) or < 2000 ng/mL, whichever was lower.
Time Frame: From first date of response and first date of loss of response or death (maximum 416 days)
Population: Enrolled-06 population included participants previously enrolled and treated in Study NI-0501-06 (participants with MAS in Still's disease) who provided informed consent for participation in Study NI-0501-05 and who had at least 1 response.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Enrolled-06 Cohort
Number analyzed (Participants) | 13
days | 61.0 [9.0 to 358.0]

4. Secondary Outcome: Overall Survival (Enrolled-04 Cohort)
Description: Overall survival was defined as time from the date of the last emapalumab dose to the date of death. Participants without an event were censored at the time of last contact or 12 months after last dose (whichever came first). As some participants had their last emapalumab dose in the parent study (NI-0501-04), data from both NI-0501-05 and NI-0501-04 studies were considered for the assessment of overall survival.
  Kaplan-Meier methodology was used for estimation.
Time Frame: From the date of last of emapalumab dose to the date of death or last contact or 12 months after last dose, whichever came first (maximum 366 days)
Population: Enrolled-04 population included participants previously enrolled and treated in Study NI-0501-04 (participants with primary HLH) who provided informed consent for participation in Study NI-0501-05.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Enrolled-04 Cohort
Number analyzed (Participants) | 37
days | NA [NA to NA] — Median and Inter-Quartile Range was not reached due to low number of events.

5. Secondary Outcome: Overall Survival (Enrolled-06 Cohort)
Description: Overall survival was defined as time from the date of last emapalumab dose to the date of death. Participants without an event were censored at the time of last contact or 12 months after last dose (whichever came first). As participants in the Enrolled-06 Cohort did not receive emapalumab in the current study, data from both NI-0501-05 and NI-0501-06 studies were considered for the assessment of overall survival.
  Kaplan-Meier methodology was used for estimation.
Time Frame: as for outcome 4
Population: Enrolled-06 population included participants previously enrolled and treated in Study NI-0501-06 (participants with MAS in Still's disease) who provided informed consent for participation in Study NI-0501-05.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Enrolled-06 Cohort
Number analyzed (Participants) | 14
days | NA [NA to NA] — Median and Inter-Quartile Range was not reached due to no event.

6. Secondary Outcome: Percentage of Participants Who Achieved Engraftment (Enrolled-04 Cohort)
Description: For participants who underwent HSCT either in parent study (NI-0501-04) or current study (NI-0501-05), engraftment rate was based on the number of participants experiencing primary or secondary graft failure (blood stem cell transplant failure, engraft failure, or transplant dysfunction), as reported as an adverse event.
Time Frame: From HSCT up to 12 months
Population: Enrolled-04 population included participants previously enrolled and treated in Study NI-0501-04 (participants with primary HLH) who provided informed consent for participation in Study NI-0501-05 and who underwent HSCT.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enrolled-04 Cohort
Number analyzed (Participants) | 29
percentage of participants | 20.7 [9.8 to 38.4]

7. Secondary Outcome: Percentage of Participants Who Achieved Donor Chimerism (Enrolled-04 Cohort)
Description: For participants who underwent HSCT, achievement of donor chimerism was considered based on donor chimerism in peripheral blood completed, that is, donor cells >95%.
Time Frame: From HSCT to 12 months
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enrolled-04 Cohort
Number analyzed (Participants) | 29
percentage of participants | 72.4 [54.3 to 85.3]

8. Secondary Outcome: Percentage of Participants With Graft-versus-host-disease (Enrolled-04 Cohort)
Description: Occurrence of graft-versus-host-disease, reported in Study NI-0501-05 as an AE.
Time Frame: From HSCT to 12 months
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enrolled-04 Cohort
Number analyzed (Participants) | 29
percentage of participants | 24.1 [12.2 to 42.1]

9. Secondary Outcome: MAS Activity Level as Assessed by Visual Analogue Scale (Enrolled-06 Cohort)
Description: MAS activity was monitored using a visual analogue scale ranging from 0 to 10 with a higher score indicted higher disease activity.
Time Frame: Baseline (first NI-0501-05 visit), Day 100, Month 12/End of Study
Population: Enrolled-06 population included participants previously enrolled and treated in Study NI-0501-06 (participants with MAS in Still's disease) who provided informed consent for participation in Study NI-0501-05 and had available data for MAS activity.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enrolled-06 Cohort
Number analyzed (Participants) | 13
score on a scale
  Baseline | 0.0 (0.0)
  Day 100: number analyzed (Participants) | 12
  Day 100 | 0.0 (0.0)
  Month 12/End of Study | 0.2 (0.48)

10. Secondary Outcome: Circulating Emapalumab Level (Enrolled-04 Cohort)
Description: Circulating Emapalumab level in Enrolled-04 Cohort who continued to receive treatment with emapalumab in the current study (NI-0501-05).
Time Frame: First infusion day (infusion duration: 1-2 hours) in Study NI-0501-05, last infusion day (infusion Day 188), 12 months post-transplant
Population: Enrolled-04 population included participants previously enrolled and treated in Study NI-0501-04 (participants with primary HLH) who provided informed consent for participation in Study NI-0501-05 and who had data available for specified timepoints. Circulating emapalumab level post-transplant included participants who had HSCT and data available at 12 months post-HSCT (Samples were not to be taken once it had been determined that emapalumab was below measurable level of 62.5 µg/L).
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Enrolled-04 Cohort
Number analyzed (Participants) | 22
µg/L
  Infusion Day 1 | 165148.4 (175057.98)
  Infusion Day 188: number analyzed (Participants) | 2
  Infusion Day 188 | 157849.0 (66180.28)
  12 months post-transplant: number analyzed (Participants) | 12
  12 months post-transplant | 80.5 (43.52)

11. Secondary Outcome: Circulating Emapalumab Level (Enrolled-06 Cohort)
Time Frame: Baseline (first NI-0501-05 visit), Day 100, Month 6
Population: Enrolled-06 population included participants previously enrolled and treated in Study NI-0501-06 (participants with MAS in Still's disease) who provided informed consent for participation in Study NI-0501-05 and had available data at specified timepoints (Samples were not to be taken once it had been determined that emapalumab was below measurable level of 62.5 µg/L).
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Enrolled-06 Cohort
Number analyzed (Participants) | 12
µg/L
  Baseline | 20968.0 (18226.14)
  Day 100: number analyzed (Participants) | 10
  Day 100 | 8515.3 (6814.50)
  Month 6: number analyzed (Participants) | 8
  Month 6 | 1628.5 (1427.46)

12. Secondary Outcome: Total Human Interferon Gamma Levels (Enrolled-04 Cohort)
Time Frame: First infusion day (infusion duration: 1-2 hours) in Study NI-0501-05, Day 100 post-transplant, 12 months post-transplant
Population: Enrolled-04 population included participants previously enrolled and treated in Study NI-0501-04 (participants with primary HLH) who provided informed consent for participation in Study NI-0501-05 and who had data available for specified timepoints. Total human interferon gamma levels post-transplant included participants who underwent HSCT and data available at Day 100 and 12 months post-HSCT.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Enrolled-04 Cohort
Number analyzed (Participants) | 24
ng/L
  Infusion Day 1: number analyzed (Participants) | 11
  Infusion Day 1 | 5290.4 (4992.27)
  Day 100 post-transplant: number analyzed (Participants) | 23
  Day 100 post-transplant | 3613.6 (6052.31)
  12 months post-transplant | 447.4 (1096.99)

13. Secondary Outcome: Total Human Interferon Gamma Levels (Enrolled-06 Cohort)
Time Frame: Baseline (first NI-0501-05 visit), Day 100, Month 12/End of Study
Population: Enrolled-06 population included participants previously enrolled and treated in Study NI-0501-06 (participants with MAS in Still's disease) who provided informed consent for participation in Study NI-0501-05 and had available data at specified timepoints.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Enrolled-06 Cohort
Number analyzed (Participants) | 13
ng/L
  Baseline | 5544.3 (8285.12)
  Day 100: number analyzed (Participants) | 12
  Day 100 | 2958.7 (6762.62)
  Month 12/End of Study: number analyzed (Participants) | 9
  Month 12/End of Study | 1111.0 (1311.04)

14. Secondary Outcome: Number of Participants With Anti-drug Antibody
Time Frame: From enrolment up to 12 months post-transplant or last emapalumab infusion (maximum 639 days)
Population: Participants who previously received treatment in a parent study (NI-0501-04 or NI-0501-06) or under CU and who provided informed consent for participation in Study NI-0501-05. Number of participants analysed included participants who had available data for anti-drug antibody.
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled-04 Cohort | Enrolled-06 Cohort | Enrolled-CU Cohort
Number analyzed (Participants) | 32 | 14 | 7
Participants | 1 | 3 | 0

ADVERSE EVENTS:
Time Frame: From the date of enrollment in this study up to 1 year either after HSCT or after the last administration of emapalumab (maximum duration: 639 days)
Description: Participants who previously received treatment in a parent study (NI-0501-04 or NI-0501-06) or under CU and who provided informed consent for participation in Study NI-0501-05.
Arm/Group | Enrolled-04 Cohort | Enrolled-06 Cohort | Enrolled-CU Cohort
All-Cause Mortality (participants affected / at risk) | 9/37 | 0/14 | 2/7
Serious Adverse Events (participants affected / at risk) | 28/37 | 3/14 | 6/7
Other Adverse Events (participants affected / at risk) | 37/37 | 11/14 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enrolled-04 Cohort (N=37) | Enrolled-06 Cohort (N=14) | Enrolled-CU Cohort (N=7)
Coombs positive haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0
Right ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Eye movement disorder (Eye disorders) | 1 | 0 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 6 | 0 | 0
Condition aggravated (General disorders) | 5 | 1 | 2
Multiple organ dysfunction syndrome (General disorders) | 2 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Acute graft versus host disease in intestine (Immune system disorders) | 2 | 0 | 0
Engraftment syndrome (Immune system disorders) | 2 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Septic shock (Infections and infestations) | 4 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 3 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 2 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 2 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Enterococcal infection (Infections and infestations) | 1 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Gianotti-Crosti syndrome (Infections and infestations) | 1 | 0 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 1 | 0 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Engraft failure (Injury, poisoning and procedural complications) | 2 | 0 | 0
Blood stem cell transplant failure (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neurological decompensation (Nervous system disorders) | 1 | 0 | 0
Subdural hygroma (Nervous system disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Shock (Vascular disorders) | 1 | 0 | 0
Still's disease (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Device breakage (Product Issues) | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enrolled-04 Cohort (N=37) | Enrolled-06 Cohort (N=14) | Enrolled-CU Cohort (N=7)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Macrocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 6 | 0 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 1
Cyanosis (Cardiac disorders) | 1 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 0
Right ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Eye movement disorder (Eye disorders) | 1 | 0 | 0
Maculopathy (Eye disorders) | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 1 | 0 | 0
Retinal disorder (Eye disorders) | 1 | 0 | 0
Retinal ischaemia (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 11 | 0 | 0
Vomiting (Gastrointestinal disorders) | 9 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 0 | 0
Oral pain (Gastrointestinal disorders) | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastric mucosa erythema (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Oral mucosal discolouration (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 17 | 1 | 1
Mucosal inflammation (General disorders) | 7 | 0 | 0
Condition aggravated (General disorders) | 5 | 0 | 1
Oedema (General disorders) | 2 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0
Complication associated with device (General disorders) | 1 | 0 | 0
Complication of device insertion (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Fibrosis (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Swelling face (General disorders) | 1 | 0 | 0
Visceral pain (General disorders) | 1 | 0 | 0
Xerosis (General disorders) | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 1 | 0 | 0
Graft versus host disease in skin (Immune system disorders) | 4 | 0 | 1
Allergy to immunoglobulin therapy (Immune system disorders) | 2 | 0 | 0
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 2 | 0 | 0
Graft versus host disease in liver (Immune system disorders) | 2 | 0 | 0
Acute graft versus host disease in skin (Immune system disorders) | 1 | 0 | 0
Bacille Calmette-Guerin scar reactivation (Immune system disorders) | 1 | 0 | 0
Engraftment syndrome (Immune system disorders) | 1 | 0 | 0
Graft versus host disease (Immune system disorders) | 1 | 0 | 1
Cytomegalovirus infection reactivation (Infections and infestations) | 5 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 3 | 0 | 0
Rhinitis (Infections and infestations) | 3 | 0 | 2
Staphylococcal bacteraemia (Infections and infestations) | 3 | 0 | 0
Adenovirus infection (Infections and infestations) | 2 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 2 | 0 | 0
Gastroenteritis adenovirus (Infections and infestations) | 2 | 0 | 0
Otitis externa (Infections and infestations) | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
BK virus infection (Infections and infestations) | 1 | 0 | 0
Bacillus bacteraemia (Infections and infestations) | 1 | 0 | 0
Croup infectious (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0
Epstein-Barr viraemia (Infections and infestations) | 1 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0 | 0
Herpes simplex gastritis (Infections and infestations) | 1 | 0 | 0
Human herpesvirus 6 infection reactivation (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0 | 0
Meningitis enterococcal (Infections and infestations) | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 1
Rhinovirus infection (Infections and infestations) | 1 | 1 | 0
Serratia bacteraemia (Infections and infestations) | 1 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 1 | 0 | 0
Skin bacterial infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Urinary tract infection viral (Infections and infestations) | 1 | 0 | 0
Viral haemorrhagic cystitis (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 4 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood stem cell transplant failure (Injury, poisoning and procedural complications) | 1 | 0 | 1
Burns first degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Engraft failure (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Transplant dysfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Unintentional medical device removal (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Transaminases increased (Investigations) | 4 | 0 | 0
Adenovirus test positive (Investigations) | 2 | 0 | 0
BK polyomavirus test positive (Investigations) | 2 | 0 | 0
Human rhinovirus test positive (Investigations) | 2 | 0 | 0
Roseolovirus test positive (Investigations) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Atypical mycobacterium test positive (Investigations) | 1 | 0 | 0
Blood albumin decreased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Blood electrolytes abnormal (Investigations) | 1 | 0 | 0
Blood immunoglobulin G decreased (Investigations) | 1 | 0 | 0
Campylobacter test positive (Investigations) | 1 | 0 | 0
Clostridium test positive (Investigations) | 1 | 0 | 0
Cytomegalovirus test positive (Investigations) | 1 | 0 | 0
Herpes simplex test positive (Investigations) | 1 | 0 | 0
Mycobacterium test positive (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Norovirus test positive (Investigations) | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Pseudomonas test positive (Investigations) | 1 | 0 | 0
Respirovirus test positive (Investigations) | 1 | 0 | 0
Urine output decreased (Investigations) | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Milk soy protein intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0
Poor feeding infant (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Growth failure (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 0
Somnolence (Nervous system disorders) | 2 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Hypotonia (Nervous system disorders) | 1 | 0 | 0
Nystagmus (Nervous system disorders) | 1 | 0 | 0
Opisthotonus (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Subdural effusion (Nervous system disorders) | 1 | 0 | 0
Irritability (Psychiatric disorders) | 4 | 0 | 0
Agitation (Psychiatric disorders) | 2 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Separation anxiety disorder (Psychiatric disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 3 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0
Scrotal swelling (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal flaring (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 5 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 9 | 0 | 1
Hypotension (Vascular disorders) | 4 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 0
Hyperaemia (Vascular disorders) | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 2 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 1 | 0
Cestode infection (Infections and infestations) | 0 | 1 | 0
Enterovirus infection (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Adverse event following immunisation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Still's disease (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sickle cell trait (Congenital, familial and genetic disorders) | 0 | 0 | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 1
Food allergy (Immune system disorders) | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 1
Enterobacter sepsis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Tracheitis (Infections and infestations) | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Torus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Acinetobacter test positive (Investigations) | 0 | 0 | 1
Candida test positive (Investigations) | 0 | 0 | 1
Klebsiella test positive (Investigations) | 0 | 0 | 1
Ubiquinone decreased (Investigations) | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertrophic osteoarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Pleocytosis (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Anuria (Renal and urinary disorders) | 0 | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communication prior to public release. The PI shall consider the comments received from the sponsor and shall delete any confidential information. The sponsor may require the delay of publication submission if it contains any patentable subject matter which requires protection.

DOCUMENTS (2):
  • Study Protocol (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/99/NCT02069899/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT02069899/SAP_001.pdf